CLINICAL TRIAL: NCT04333043
Title: Evaluation of the Hearing Aids Efficacy in Elderly Subjects: a Protocol for Multiparametric Longitudinal Study
Brief Title: Hearing Aids Use in Elderly: Efficacy in Speech Perception and in Health-related Quality of Life
Status: Completed | Type: Observational
Sponsor: Azienda Unita Sanitaria Locale di Piacenza (Other)
Responsible Party: Principal Investigator, Sara Ghiselli, Principal investigator, MD, Head of Otolaryngology, PhD student, Azienda Unita Sanitaria Locale di Piacenza
Other Study IDs: HA Elderly 2020
Record Dates: First submitted 2020-03-26; First posted 2020-04-03 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Hearing Loss, Age-Related
MeSH Terms: conditions — Presbycusis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hearing Aids: Hearing Aids use
  Interventions: Diagnostic Test: audiological test, cognitive questionnaires

INTERVENTIONS:
Diagnostic Test: audiological test, cognitive questionnaires — administration of cognitive and quality of life questionnaires and audiological test

SUMMARY:
Background: Prevalence of hearing loss increases over age; its estimated prevalence is 40-50% in people older than 75 years. Recent studies agree that modification in the hearing threshold contributes to deterioration in sociality, sensitivity, cognition, and quality of life of the elderly subjects.

Our study objective is to verify if rehabilitation with first time applied Hearing Aids (HA) in a cohort of old people with hearing impairment improves over time speech perception in a noisy environment and the overall health-related quality of life.

Methods: The monocentric, prospective, repeated measures, single-subject, clinical observational study will accrue 100 elderly, first-time HA recipients (≥ 65 years). The evaluation protocol is designed to analyze changes on specific measurement tools a year after the first HA fitting in comparison to the evaluation before HA usage.

Evaluations will consist of multiparametric details collected through self-report questionnaires completed by the recipients and a series of commonly used audiometric measures and geriatric assessment tools. The primary indicator of changes in speech perception in noise will be the OLSA test whereas the indicator of changes in overall quality of life will be the AQoL and HHEI questionnaires. Montreal Cognitive Assessment (MoCA) will help us to verify the cognitive state of the subjects. This questionnaire will allow us to exclude a reduction of the cognitive abilities over time.

Discussion: The protocol is designed to make use of measurement tools that have already been applied to the hearing-impaired population in order to compare the effects of HA rehabilitation in the elderly immediately before their first HA usage (Pre) and after gaining 1 year of experience (Post). The broad approach will lead to a greater understanding of how useful hearing influences the quality of life in elderly individuals, and thus improves potentials for healthy aging. Outcomes will be described and analyzed in detail.

DETAILED DESCRIPTION:
This study wants to identify significant improvement in speech recognition in noise in elderly patients (>= 65 years) that use HA for the first time and the correlations between the use of the HA and quality of life and cognitive status in elderly patients.

This is a repeated measure, single-subject, prospective observational study. No additional intervention is applied to population of HA recipients. Study subjects who use for the first time unilateral or bilateral hearing aids will be included. Eligible participants are consecutively identified on the HA registry of the Local Unit of the National Health System (NHS). Italian NHS is a welfare system which funds totally or partially the HA costs in selected patients.

An approximate number of 100 individuals will be included. The study design is monocentric and it is conducted at the outpatient service of the ENT Department of the "Saliceto" Hospital.

The test includes language-appropriate materials relative to the participating HA recipient.

The evaluation protocol is designed to coincide with routine clinical visits. Each subject is assessed with the full test-battery and questionnaires that are repeated at each of the two visits: one before the HA fitting (Pre) and one after one year of HA use (Post).

Subjects are enrolled in the clinical investigation only after signing the Patient Informed Consent Form prior to the first assessment (baseline, t0).

During the first assessment (Pre) are carried out this procedures: otoscopy and cleaning of the external auditory canal,- unaided pure tone audiometry, unaided speech audiometry in quiet, Italian version of Oldenburg Satztest (OLSA test) and Montreal Cognitive Assessment (MOCA), Hearing Handicap Inventory in the Elderly Screening test (HHIE-S) and Assessment of Quality of Life (AQoL) questionnaires.

During the second assessment (Post) are carried out: otoscopy and cleaning of the external auditory canal, test of the HA functioning, unaided pure tone audiometry, aided speech audiometry in quiet, Italian version of OLSA test and MOCA, HHIE-S, AQoL and International Outcome Inventory for Hearing Aids (IOI-HA) questionnaires.

The maximum administration time for completion of all measures is estimated to be approximately one hour of which 30 minutes are dedicated to standard self-report forms completed by the HA recipient.

In addition to general healthcare and patient-profile data, a selection of observational clinical assessment tools has been chosen for repeated evaluations to reflect changes in the hearing aid benefit and the overall health status of the elderly individual at post-HA use. These tools are commonly used in audiology and/or geriatric practices and are administered in the appropriate language. All questionnaires are validated for the Italian language.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 65 years
* First use of unilateral or bilateral HA
* HA partially or totally funded by the National Health System
* Willingness to participate in and to comply with all study procedures
* Fluency in languages used to assess clinical performance
* Able to decide on study participation personally, and independently sign their consent

Exclusion Criteria:

* Unilateral hearing loss
* Previous use of HA
* Significantly/severely dependent or fragile
* Unable to provide consent personally
* Unable to complete questionnaires for self-assessment independently
* Significant comorbidities preventing study participation (e.g. blindness, immobility or in a wheelchair, severe aphasia, and other)
* Unrealistic expectations on the part of the subject regarding the possible benefits, risks and limitations inherent to the procedure and prosthetic device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study subjects who use for the first time unilateral or bilateral hearing aids will be included. Eligible participants are consecutively identified on the HA registry of the Local Unit of the National Health System (NHS). Italian NHS is a welfare system which funds totally or partially the HA costs in selected patients.
  Subjects are > = 65 years old people using unilateral or bilateral HA for the first time. According to local NHS threshold-criteria for funding adult's HAs, patients' best ear must have a Pure-Tone Average >= 45 dB HL. Subjects are enrolled in the clinical investigation only after signing the Patient Informed Consent Form prior to the first assessment (baseline, t0). An approximate number of 100 individuals will be included.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-02-07 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Improvement in speech recognition in noise with audiometrical test | up to 12 months
  The primary aim is to identify significant improvement in speech recognition in noise in elderly patients (>= 65 years) that use Hearing Aids for the first time.
  To verify this aim, our patients are subject to audiometric tests in quiet conditions.
  Audiometric test include standard threshold measures for frequencies 250-4000 Hz (pure tone audiogram) and speech discrimination (speech audiometry).
  Normal hearing patients show an average threshold less than 30 dB in the pure tone audiogram.
  Speech audiometry shows the Speech Reception Threshold (SRT), defined as the level of speech corresponding to 50% of correct answers. Normal hearing patients show a SRT at 30 dB.
Improvement in speech recognition in noise with OLSA test | up to 12 months
  The primary aim is to identify significant improvement in speech recognition in noise in elderly patients (>= 65 years) that use Hearing Aids for the first time.
  The primary aim is to identify significant improvement in speech recognition in noise in elderly patients (>= 65 years) that use Hearing Aids for the first time.
  To verify this aim, our patients are subject to audiometric tests in noise condition.
  The audiometric test in noise condition is a speech adaptive audiometry: Italian version of Oldenburg Satztest (OLSA test). The test is conducted using a closed-set response format.
  Puglisi et al. (2015) described the reference ranges and standard deviations of the OLSA test for the Italian language. The cutoff of the SNR dB (SRT) among the elderly was set to - 0.4 dB based on a reference mean level of -6.7 plus 2 standard deviations. Lower scores underlines a better performances.

SECONDARY OUTCOMES:
Hearing Aids and quality of life with AQoL-8D questionnaire | up to 12 months
  The secondary aim is to process the correlations between the use of the HA and quality of life in elderly.
  To verify this aim, our patients are subject to this questionnaire: Assessment of Quality of Life (AQoL).
  The AQoL-8D consists of five psychosocial and three physical dimension. The AQoL includes 35 items with 5 possible answers; this questionnaire does not have a score scale.
Hearing Aids and cognitive skills with MOCA questionnaire | up to 12 months
  The secondary aim is to process the correlations between the use of the HA and cognitive status in elderly.
  To verify this aim, our patients are subject to this questionnaire: Montreal Cognitive Assessment (MoCA).
  MoCA detects cognitive impairment. It consisting of 12 subtasks. The total score ranges from 0 (worst performance) to 30 (best performance). The presence of mild cognitive dysfunction is suspected when the final score is less than 26.
Hearing Aids and cognitive skills and quality of life with IOI-HA questionnaire | up to 12 months
  The secondary aim is to process the correlations between the use of the HA and quality of life and cognitive status in elderly.
  To verify this aim, our patients are subject to this questionnaire: International Outcome Inventory for Hearing Aids (IOI-HA).
  IOI-HA quantifies the satisfaction of hearing aid users. The IOI-HA contains seven domains used to subjectively evaluate the results of the HA under the following parameters: (1) time for which HA have been used; (2) benefit; (3) residual limitation in daily life activities; (4) satisfaction; (5) residual restrictions to participation; (6) impact on other people; and (7) quality of life.
  The answers to each question range from poor performance (1) to best performance (5).
  A high score is an indication of good outcome in aided conditions.
Hearing Aids and cognitive skills with HHIE-S questionnaire | up to 12 months
  The secondary aim is to process the correlations between the use of the HA and cognitive status in elderly.
  To verify this aim, our patients are subject to this questionnaire: Hearing Handicap Inventory for the Elderly Screening Version (HHIE-S).
  HHIE-S assess the effects of hearing impairment on emotional and social adjustment in everyday life.
  This test contains a 10-item questionnaire. The answers to each question range from poor performance (0) to best performance (4). A low HHIE-S total score indicates less perceived difficulties.

CONTACTS AND LOCATIONS:
Overall Officials: Domenico Cuda, MD, Principal Investigator — Ospedale Guglielmo da Saliceto, Piacenza
Locations (1):
- Ospedale Guglielmo da Saliceto- ENT Department, Piacenza, PC, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ghiselli S, Soncini A, Fabrizi E, Salsi D, Cuda D. Factors correlated with hearing aids adherence in older adults: a prospective controlled study. J Int Med Res. 2024 Jun;52(6):3000605241232549. doi: 10.1177/03000605241232549. PMID 38861681
- [Derived] Cuda D, Ghiselli S, Murri A. Evaluation of the efficacy of hearing aids in older adults: a multiparametric longitudinal study protocol. BMC Geriatr. 2021 Feb 5;21(1):107. doi: 10.1186/s12877-021-02033-z. PMID 33581722